CLINICAL TRIAL: NCT01496456
Title: Radiographic Progression of Infiltrated Caries Lesions In-vivo
Acronym: ICON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Principal Investigator, Mathilde Peters, DMD, PhD, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG#N010508; 10-PAF03721 (Other: U-Michigan)
Record Dates: First submitted 2011-12-09; First posted 2011-12-21 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Dental Caries
Keywords: Dental caries; Proximal surfaces; Posterior teeth; Carious lesions; Tooth diseases; Preventive therapy
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preventative measures (Placebo Comparator): Caries management by preventative measures of oral hygiene instruction, diet counseling and fluoride supplementation
  Interventions: Behavioral: Caries management
- Lesion infiltration (Active Comparator): Resin infiltration of caries lesion in addition to caries management by preventative measures of oral hygiene instruction, diet counseling and fluoride supplementation
  Interventions: Device: Resin infiltration; Behavioral: Caries management

INTERVENTIONS:
Device: Resin infiltration — Split-mouth design (at least two lesions per patient): Treatment of one caries lesion with resin infiltration therapy
  Other Names: ICON (DMG, Germany)
  Arms: Lesion infiltration
Behavioral: Caries management — Split-mouth design (at least two lesions per patient). Baseline preventative caries management: dietary and behavioral modification, and over-the-counter fluoride supplements
  Other Names: Home use of over-the-counter oral health products

SUMMARY:
This study is investigating the efficacy of caries lesion infiltration therapy as compared to the current preventative approach for early caries lesions.

DETAILED DESCRIPTION:
A 3-year longitudinal, prospective, randomized control clinical trial (RCT) is designed incorporating a split-mouth intra-oral design. Young volunteers (14-35 years old) with at least two early lesions in posterior teeth will be enrolled into this clinical trial to evaluate the clinical effectiveness of arresting lesion progression by infiltrating the lesions. The infiltration protocol included application of on-market materials and applicators, and was performed in one session.

ELIGIBILITY:
Inclusion Criteria:

* 14-35 year old subjects
* decayed-missing-filled permanent teeth (DMFT) ≥ 3
* having at least two early caries lesions in approximal posterior tooth surfaces
* lesion visible on radiograph

Exclusion Criteria:

* Current participation in another clinical study
* Medically compromised subjects
* Hyposalivation
* Pregnancy
* Allergic to methylmethacrylates
* Allergic to latex
* Symptomatic teeth

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Chair — University of Michigan
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peters MC, Tuzzio F, Nedley M, Davis W, Bayne SC. Resin Infiltration Effects In A Caries-Active Environment. J Dent Res 92(Spec Iss A):377, 2013.
- [Result] Resin infiltration effects in a caries-active environment. J Calif Dent Assoc. 2014 Jun;42(6):372. No abstract available. PMID 25080756
- [Result] Peters MC, Bula A, Nedley M, Davis W, Bayne SC. Efficacy of Resin Infiltration in High Caries-Active Environment -- 3YR Results. J Dent Res 93(Spec Iss B): 1017, 2014.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was not as expected and halted after one year. Local options to enhance patient accrual were exhausted. The total patient pool was small, but of sufficient scientific value to continue and complete the study.
Pre-assignment Details: Paired, split-mouth study design: Each patient received at least 1 pair of 2 treatments (one of each arm). Eligible tooth pairs selected for similarity. Random allocation of treatment to study teeth of each tooth pair.
Groups:
- Lesion Infiltration and Preventative Management Only: Paired split-mouth study: both arms (arm A and arm B) were applied in same patient (2 study teeth).
  A) Resin infiltration therapy in addition to SOC Preventative caries management B) SOC Preventative caries management only.
  --- Standard Of Care (SOC) Baseline preventative caries management included dietary and behavioral modification, and over-the-counter (OTC) fluoride supplements.
Period: Overall Study
Arm/Group | Lesion Infiltration and Preventative Management Only
Started | 17
Baseline | 16 (Baseline group started with 16 patients.)
1-yr Recall | 12
2-yr Recall | 10
3-yr Final Recall | 9
Completed | 9
Not Completed | 8
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: Enrolled: 17 patients; 1 patient was not treated according to protocol. Baseline: 16 patients with 22 tooth pairs.
Groups:
- Lesion Infiltration and Preventative Management Only: Paired split-mouth study: both arms in same patient (2 study teeth). A) Resin infiltration therapy in addition to preventative caries management B) Preventative caries management only
  SOC Baseline preventative caries management: dietary and behavioral modification, and OTC fluoride supplements
Arm/Group | Lesion Infiltration and Preventative Management Only
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions Showing Radiographic Progression as Measured by Lesion Size (Continuous)
Description: Pairwise radiographic assessment of lesion progression: combined visual assessment (PWA) and digital subtraction radiography (DSR).
Time Frame: Baseline through 3 years
Population: Pairwise assessment: visual (PWA) + digital subtraction radiography (DSR).
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Lesion Infiltration: Resin infiltration of caries lesion in addition to SOC caries management by preventative measures.
- Preventative Measures: SOC Caries management by preventative measures only.
Arm/Group | Lesion Infiltration | Preventative Measures
Number analyzed (Participants) | 9 | 9
Number analyzed (Lesions) | 13 | 13
Lesions | 2 | 11
Statistical Analysis 1: Comparison: Lesion Infiltration vs Preventative Measures; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Ordinal logistic regression, controlled for baseline lesion size and for correlation among pairs of teeth using the GEE method

2. Secondary Outcome: Number of Lesions Showing Radiographic Progression as Measured by Lesion Depth Categories
Description: Radiographic assessment of lesion depth category (R1-R5) by single radiograph assessment (SRA).
Time Frame: Baseline through 3 years
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Preventative Measures: Caries management by preventative measures only: oral hygiene instruction, diet counseling and fluoride supplementation
  Baseline SOC preventative caries management: dietary and behavioral modification, and OTC-fluoride supplements
Arm/Group | Lesion Infiltration | Preventative Measures
Number analyzed (Participants) | 9 | 9
Number analyzed (Lesions) | 13 | 13
Lesions | 2 | 9
Statistical Analysis 1: Comparison: Lesion Infiltration vs Preventative Measures; Test type: Superiority or Other; p = 0.045, Regression, Logistic; Ordinal logistic regression, controlled for correlation among pairs of teeth using the GEE method

3. Secondary Outcome: Lesion Survival After 3 Years
Description: Discrete time survival analysis of time to first lesion progression.
Time Frame: 3 years
Population: Radiographic lesion increase by PWA+DSR. A tooth was included up until the time the lesion first increased.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Lesion Infiltration | Preventative Measures
Number analyzed (Participants) | 13 | 13
Number analyzed (Lesions) | 18 | 18
Lesions | 11 | 3
Statistical Analysis 1: Comparison: Lesion Infiltration vs Preventative Measures; Test type: Superiority or Other; p = 0.0077, Discreet Time Survival Analysis; Controlled for correlation among tooth pairs (GEE model)

ADVERSE EVENTS:
Time Frame: Baseline through 3 years
Groups:
- Lesion Infiltration: Resin infiltration of caries lesion in addition to SOC caries management by preventative measures
  SOC Baseline preventative caries management: dietary and behavioral modification, and OTC-fluoride supplements
- Preventative Measures: Caries management by preventative measures only
  SOC Baseline preventative caries management: dietary and behavioral modification, and OTC-fluoride supplements
Arm/Group | Lesion Infiltration | Preventative Measures
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes